CLINICAL TRIAL: NCT05306782
Title: The Treatment of Persistent Developmental Stuttering: Shaping of Motor Neural Functioning to Improve Fluency
Brief Title: Shaping Motor Neural Functioning of Developmental Stuttering to Improve Fluency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Pierpaolo Busan, Principal Investigator, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: GR-2018-12366027
Record Dates: First submitted 2022-02-26; First posted 2022-04-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Stuttering
Keywords: Developmental Stuttering; Neuromodulation; transcranial Electrical Stimulation; Speech Fluency; Motor Networks
MeSH Terms: conditions — Stuttering | interventions — Transcranial Direct Current Stimulation; Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomly assigned to "real" neuromodulation or to "sham" modulation (in addition to speech therapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial Random Noise Stimulation (Experimental): Transcranial Random Noise Stimulation (1.5 mA, High Frequency) administered by using surface scalp electrodes (20 minutes, initial part of the session) in correspondence of associative motor regions, during speech therapy sessions (45 minutes).
  Interventions: Device: transcranial Electrical Stimulation; Behavioral: Speech Therapy
- Transcranial Direct Current Stimulation (Experimental): Transcranial Direct Current Stimulation (1.5 mA, anodal) administered by using surface scalp electrodes (20 minutes, initial part of the session) in correspondence of associative motor regions, during speech therapy sessions (45 minutes).
  Interventions: Device: transcranial Electrical Stimulation; Behavioral: Speech Therapy
- Sham Direct Current/Random Noise Stimulation (Sham Comparator): Sham stimulation administered by using surface scalp electrodes (20 minutes, initial part of the session) in correspondence of associative motor regions, during speech therapy sessions (45 minutes).
  Interventions: Device: transcranial Electrical Stimulation; Behavioral: Speech Therapy

INTERVENTIONS:
Device: transcranial Electrical Stimulation — transcranial Random Noise Stimulation, transcranial Direct Current Stimulation, or Sham are administered (by means of surface electrodes) on associative motor regions during speech therapy sessions (20 minutes, in the initial part of the sessions; 1.5 mA).
Behavioral: Speech Therapy — Speech Therapy is associated to transcranial electrical stimulation or sham, during stimulation sessions. Total duration of the single session: 45 minutes

SUMMARY:
Developmental stuttering (DS) is a motor/speech disorder, characterized by specific alterations in the functioning of brain circuits. Non-invasive brain stimulation may be useful to shape the altered functioning and connectivity of these systems. As a consequence, this project aims to expand the neurophysiological understanding of DS, evaluating effects of transcranial electrical stimulation (tES) on speech fluency and brain functioning of adults with persistent DS. This project will provide high-impact insights into the functioning of DS neural system, also proposing innovative and/or personalized rehabilitation.

DETAILED DESCRIPTION:
Investigators will evaluate the effect of different tES protocols targeting motor associative regions (about 10 "consecutive" stimulation sessions, in different days; tES will be compared to sham stimulation), in association with "canonical" speech therapy. About 30 right-handed adults with idiopathic and persistent DS since childhood will be recruited (age 18-59 years; please see below for inlusion/exclusion criteria). Participants will be subdivided in three groups (in association to speech therapy): two groups will undergo transcranial random noise stimulation or transcranial direct current stimulation, while the third group will undergo sham (placebo) stimulation . Effects will be assessed by measuring stuttering severity (i.e. objective evaluation of stuttering), behavioral/cognitive scales (i.e. subjective evaluation of stuttering), as well as a series of neurophysiological indexes useful to evaluate brain functioning and connectivity (e.g. TMS[transcranial magnetic stimulation]-induced motor/evoked potentials and EEG brain activity). Evaluations will be realized before the start of the tES protocols, as well as at the end of the cycles. Follow-up evaluations (starting from about 6 weeks after completion of stimulation sessions) are also foreseen after the end of the treatments.

ELIGIBILITY:
(main) Inclusion Criteria:

-Right-handed adults with idiopathic, persistent DS since childhood

(main) Exclusion Criteria:

* Contraindications to non-invasive brain stimulation;
* Currently assumption of drugs acting on the Central Nervous System;
* Presence of overt neurological/psychiatric/medical conditions or overt comorbidities (e.g. obsessive-compulsive disorder).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Speech Fluency and Stuttering Severity (change from baseline) | Evaluated immediately after the end of treatments
  Utilization of (objective) scales to evaluate stuttering severity and speech fluency (Stuttering Severity Instrument [range 0-56; higher values indicate higher numbers of dysfluencies])
TMS-induced (Motor) Evoked Potentials (change from baseline) | Evaluated immediately after the end of treatments
  Utilization of Transcranial Magnetic Stimulation to evaluate excitability (and reactivity) of motor cortex
EEG (change from baseline) | Evaluated immediately after the end of treatments
  Utilization of EEG to evaluate brain functioning and brain connectivity (delta, theta, alpha, beta, and gamma activity)

SECONDARY OUTCOMES:
Stuttering Severity (subjective perception) (change from baseline) | Evaluated immediately after the end of treatments
  Utilization of (subjective) scales to evaluate stuttering severity/speech fluency (e.g. Premonitory Awareness in Stuttering Scale [range 0-42; higher values indicate higher "invasiveness" of stuttering with respect to quality of life])
Stuttering Severity (subjective perception) (change from baseline) | Evaluated about 6 weeks after the end of treatments
  Utilization of (subjective) scales to evaluate stuttering severity/speech fluency (e.g. Premonitory Awareness in Stuttering Scale [range 0-42; higher values indicate higher "invasiveness" of stuttering with respect to quality of life])
Speech Fluency and Stuttering Severity (change from baseline) | Evaluated about 6 weeks after the end of treatments
  Utilization of (objective) scales to evaluate stuttering severity and speech fluency (Stuttering Severity Instrument [range 0-56; higher values indicate higher numbers of dysfluencies])
TMS-induced (Motor) Evoked Potentials (change from baseline) | Evaluated about 6 weeks after the end of treatments
  Utilization of Transcranial Magnetic Stimulation to evaluate excitability (and reactivity) of motor cortex
EEG (change from baseline) | Evaluated about 6 weeks after the end of treatments
  Utilization of EEG to evaluate brain functioning and brain connectivity (delta, theta, alpha, beta, and gamma activity)
Cognitive/behavioral indexes (associated with stuttering) (change from baseline) | Evaluated immediately after the end of treatments
  Utilization of (subjective) scales to evaluate cognitive/behavioral reactions (e.g. Beck Depression Inventory [range 0-63; higher values indicate higher presence of depressive symptoms])
Cognitive/behavioral indexes (associated with stuttering) (change from baseline) | Evaluated about 6 weeks after the end of treatments
  Utilization of (subjective) scales to evaluate cognitive/behavioral reactions (e.g. Beck Depression Inventory [range 0-63; higher values indicate higher presence of depressive symptoms])

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Busan, Dr., Principal Investigator — IRCCS Ospedale San Camillo s.r.l.
Locations (1):
- IRCCS Ospedale San Camillo, Venice, Italy

IPD SHARING:
Plan to Share IPD: No